CLINICAL TRIAL: NCT03752606
Title: Does Intraoperative Application of TachoSil Reduce the Number of Lymphocele After Pelvic Lymphadenectomy?
Brief Title: Application of Tachosil During Lymphadenectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Paweł Miotła, Clinical Proffesor, Medical University of Lublin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 022018
Record Dates: First submitted 2018-11-18; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Lymphocele; Endometrial Cancer; Cervical Cancer
Keywords: lymphadenectomy; lymphocele; endometrial cancer; cervical cancer
MeSH Terms: conditions — Lymphocele; Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A Tachosil® patch of 4.8x4.8 cm was attached to one side of the obturator fossa (study group) and the same patient constituted also control group, because no Tachosil® patch was used on the second side of lymphadenectomy. Specific drainage of the retroperitoneum was performed. Patients had to agree to participate in the study and signed informed consent at least one day before surgery. Taking into consideration the examined group the patient was allocated to, the surgeon applied either one Tachosil® patches in the study group or no Tachosil® in the control group. After placing for 4 minutes, a uniform pressure was applied to it to provide rapid haemostasis by forming a strong, fibrin clot adjacent to the tissue surface. Tachosil was placed alternately once in the left, once in the right obturator fossa, so that each of the patients participating in the study could be their own control.
Who Masked: Outcomes Assessor
Masking Description: Allocation was communicated by telephone after informed consent had been obtained and after lymphadenectomy had been completed. Outcome assessment was performed by the independent reviewers. Outcome assessors were blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACHOSIL GROUP (Active Comparator): Surgical procedures were performed by four doctors with extensive experience in oncological gynecology. A TachoSil® absorbable patch of 4.8x4.8 cm was attached, once, intraoperatively to one side of the obturator fossa (study group). Specific drainage of the retroperitoneum was performed.
  Interventions: Biological: TACHOSIL GROUP
- GROUP WITHOUT TACHOSIL (No Intervention): The same patient constituted also control group, because no TachoSil® absorbable patche was used on the second side of lymphadenectomy. Specific drainage of the retroperitoneum was performed.

INTERVENTIONS:
Biological: TACHOSIL GROUP
  Other Names: NCT01192022
  Arms: TACHOSIL GROUP

SUMMARY:
The prevention of lymphoceles was assessed using collagen patch coated with the human coagulation factors (TachoSil, Nycomed International Management GmbH, Zurich, Switzerland; NCT Number ICMJE NCT01192022; Other Study ID Numbers ICMJE TC-2402-040-SP; U1111-1130-9121 Registry Identifier: WHO) on 50 consecutive patients with endometrial and cervical cancer stages IB to II who had undergone open hysterectomy and pelvic lymphadenectomy (PL).

Methods:

Each patient was simultaneously randomized in two groups: as a control (side without Tachosil applied) and study group (side with Tachosil applied). All surgical parameters were collected and patients underwent ultrasound examination on postoperative days 1, 6, and 30, and at the end of treatment.

DETAILED DESCRIPTION:
The study was approved by the Bioethics Committee of the Medical University of Lublin, Lublin, Poland (KE-0254/276/2013). The study population consisted of 50 women undergoing pelvic lymphadenectomy for cervical and endometrial cancer and meeting the inclusion/exclusion criteria requirements. Inclusion criteria for the study included women undergoing open hysterectomy and lymphadenectomy for cervical or endometrial cancer, age between 18 and 70 years, who signed a written informed consent. Exclusion criteria included women with previously diagnosed lymph edema or disease of the lymphatic system or a known disease of the immune system. Prospective randomized clinical intervention trial of 50 open surgery during 2013-2014 at 2nd Department of Gynecology in Lublin. Women were centrally randomized by the principal investigator (TR). Surgeons allocated Tachosil for one side (left or right) after lymphadenectomy, second side was as a control side without Tachosil. Allocation was communicated by telephone after informed consent had been obtained and after lymphadenectomy had been completed. Outcome assessment was performed by the independent reviewers. Outcome assessors were blinded to the treatment allocation. The open surgery were performed as follows: in women who underwent routine pelvic lymphadenectomy, lymph node tissue was removed from the external iliac vessels, the obturator fossa, the interiliac region, and the common iliac region after identification and appropriate preparation of iliac vessels and obturator nerve. At the end of the procedure, hemostasis was checked. A Tachosil® patch of 4.8x4.8 cm was attached to one side of the obturator fossa (study group) and the same patient constituted also control group, because no Tachosil® patch was used on the second side of lymphadenectomy. Specific drainage of the retroperitoneum was performed. Patients had to agree to participate in the study and signed informed consent at least one day before surgery. Taking into consideration the examined group the patient was allocated to, the surgeon applied either one Tachosil® patches in the study group or no Tachosil® in the control group. After placing for 4 minutes, a uniform pressure was applied to it to provide rapid haemostasis by forming a strong, fibrin clot adjacent to the tissue surface. Tachosil was placed alternately once in the left, once in the right obturator fossa, so that each of the patients participating in the study could be their own control. The next step was a radical hysterectomy with adnexa. After completion of the procedure, the stump of the vagina stitching to the hollow was performed by passing the vaginal seam through the vaginal wall, the right-side sacro-uterus ligament, the right round ligament, the peritoneal uterine vesiculitis, the left round ligament, the left sacro-uterine ligament and finally the vaginal wall. This way of fixation allowed free lymphatic drainage of the retroperitoneal space. Two drains from the vicinity of the pits of the curtains were removed through the abdominal wall, which were left to the second day after surgery or longer if the volume of secretion in the drainage exceeded 40 ml per day. The urinary bladder catheter was removed on the third day after surgery and ultrasound after voiding (PVR) was evaluated. Surgical procedures were performed by four doctors with extensive experience in oncological gynecology. The surgical protocols were blinded to other researchers who controlled patients in the postoperative period. The data obtained by them were analyzed by an independent reviewer. The evaluation criteria of the study were the development of lymph cysts and their volume. Antibiotic prophylaxis was implemented according to local hospital recommendations. In addition, metronidazole was administered at a dose of 500 mg every 8 hours. i.v. for the first three days after the procedure. Patients also received small-molecule heparin at a dose of 4,000 IU from the day preceding the surgery up to 30 days after its completion. Due to the fact that lymphatic cysts usually appear 7 to 15 days after lymphadenectomy, the ultrasound examination of the presence and volume of lymphocele was performed on the 7th and 30th day after the surgery and after completing the oncological complementary treatmentThe criteria proposed by Tinelli et al. were used to define lymphocele.

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer (FIGO IA1, IA2, IB1, IB2)
* endometrial cancer (FIGO IA, IB, II)
* age between 18 and 70 years
* signed a written informed consent

Exclusion Criteria:

* lymph edema
* disease of the lymphatic system
* a known disease of the immune system

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with cervical or endometrial cancer age between 18 and 70 years signed a written informed consent
Enrollment: 50 (Actual)
Dates: Start 2013-11-29 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence and volume of lymphocele. | 1 year
  Number of participants with lymphocele as assessed by USG scan at 1,6,30 days and the drainage volume in ml with/without Tachosil assessed by USG scan at 1,2,6,30 days

SECONDARY OUTCOMES:
The incidence of lymphocele after adjuvant treatment | 1 year
  Number of participants with lymphocele as assessed by USG scan after complement adjuvant treatament

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Rechberger, Prof, Principal Investigator — IInd Department of Gynecology, Medical University of Lublin, Poland
Locations (1):
- IInd Department of Gynecology, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: from now to ongoing
Access Criteria: from the corresponding author on reasonable request.

REFERENCES:
- [Result] Tinelli A, Giorda G, Manca C, Pellegrino M, Prudenzano R, Guido M, Dell'Edera D, Malvasi A. Prevention of lymphocele in female pelvic lymphadenectomy by a collagen patch coated with the human coagulation factors: a pilot study. J Surg Oncol. 2012 Jun 15;105(8):835-40. doi: 10.1002/jso.22110. Epub 2011 Oct 10. PMID 21987409
- [Result] Tinelli A, Mynbaev OA, Tsin DA, Giorda G, Malvasi A, Guido M, Nezhat FR. Lymphocele prevention after pelvic laparoscopic lymphadenectomy by a collagen patch coated with human coagulation factors: a matched case-control study. Int J Gynecol Cancer. 2013 Jun;23(5):956-63. doi: 10.1097/IGC.0b013e31828eeea4. PMID 23574881